CLINICAL TRIAL: NCT05671523
Title: Effect Of Dry Needling On Quality Of Life In Patients With Trigger Fingers. Randomized Controlled Trail
Brief Title: Effect Of Dry Needling On Quality Of Life In Patients With Trigger Fingers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Abeer Yamany, Ph. D., principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: p.t.REC/012/003924
Record Dates: First submitted 2022-12-14; First posted 2023-01-04 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Trigger Finger Disorder
MeSH Terms: conditions — Trigger Finger Disorder | interventions — Dry Needling

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dry needling (Experimental): The patients will receive ten sessions, twice a week, for five weeks of dry needling in addition to their conventional physical therapy program (splinting and ultrasound therapy.)
  Interventions: Procedure: Dry needling; Other: conventional treatment
- conventional treatment (Active Comparator): The patients will receive conventional treatment (splinting and ultrasound therapy) for 5 weeks
  Interventions: Other: conventional treatment

INTERVENTIONS:
Procedure: Dry needling — Firstly the skin is cleaned with a piece of cotton immersed in alcohol. Then sterilized disposable thin, stainless steel needles (25 × 0.30 mm) will be inserted into the skin over the nodule in A1 pulley anatomic location. The duration of needling will be 1 minute. The needle will be inserted deeply at 45° to the level of metacarpophalangeal level to the nodule. The needle may be inserted into the tendon. This is confirmed by needle movement when the patient ﬂexes and extends the distal phalanx. The needle is withdrawn slowly until this motion ceases, and the needle tip is in the A1 pulley. This will be repeated 2 times per week for 5 weeks.
  Arms: Dry needling
Other: conventional treatment — Finger splint is designed to stabilize and immobilize a small finger joint. A wide, flat band offers comfortable pressure distribution and control. Contoured finger splint with a comfortable, close fit. The patient will use the splint at night. Can easily be adjusted to accommodate swollen digits. Suitable for a number of finger conditions.
  Therapeutic ultrasound is often used by physiotherapists to reduce pain, increase circulation and increase mobility of soft tissues. Additionally, the application of ultrasound can be helpful in the reduction of inflammation, reducing pain and the healing.

SUMMARY:
This study will be conducted to investigate the effect of dry needling on quality of life in patients with trigger finger

DETAILED DESCRIPTION:
Trigger finger (TF) is one of the most prevalent causes of hand disability and is a common cause of referral to orthopedic clinics. Trigger finger is tenosynovitis of the flexor sheaths that typically occurs in the 4th finger and thumb as a result of repetitive use. The incidence of TF is 28:100,000 per year or lifetime risk of 2.6% in the general population. It has the highest incidence being between 52 and 62 years more in women (75%). Thumb and fourth digit (ring finger) are the most commonly affected fingers.

Dry needling (DN) is a relatively new technique used by physical therapists to treat myofascial trigger points (MTrPs) and various pain syndromes. Dry needling is defined as a "skilled intervention using a thin filiform needle to penetrate the skin that stimulates myofascial TrPs, muscles, and connective tissue for the treatment of musculoskeletal pain disorders. DN has analgesic and anti-inflammatory effects, it is commonly used to relieve pain and reduce inflammation.

ELIGIBILITY:
Inclusion Criteria:

* 40 patients all have trigger fingers lasting at least 4 weeks.
* Both gender will be included
* Age of patients will be 45-75 years old
* Pain and tenderness at the position of A1 pulley.
* Nodule palpation, pain, and discomfort when flexing and extending the finger, presence of a clicking sound at the time of flexion or extension of the finger, snapping or locking of the finger.
* Willing and able to complete study procedures.

Exclusion Criteria:

* Participants with diabetes mellitus.
* History of trauma, and rheumatoid arthritis.
* Dialysis treatment.
* fingers with a history of local gouty/pyogenic disease.
* Major hand trauma and fear of needles.
* Any contraindication for deep dry needling such as anticoagulants, infections, bleeding, or psychotic conditions tumors, calcium deposits, or severe osteoarthritis.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-06-10 (Actual); Study Completion 2023-06-10 (Actual)

PRIMARY OUTCOMES:
Life quality | up to five weeks
  Quality of life will be assessed by quality of life questionnaire which is a broad concept that covers such areas as social, environmental, economic, and health satisfaction, health-related quality of life (HRQL) is less wide ranging, including mental and physical health and their consequences. Higher score denote higher quality of life and lower score denote lower quality of life. There are two methods for converting raw scores to transformed scores. The first transformation method converts score to range between 4-20,comparable with the WHOQOL-100. The second transformation method converts domain scores to a 0-100 scale.
Severity of pain | up to five weeks
  severity of pain will be assessed by visual analogue scale. Scores are based on self-reported measures of symptoms that are recorded with a single handwritten mark placed at one point along the length of a 10-cm line that represents a continuum between the two ends of the scale "no pain" on the left end (0 cm) of the scale and the "worst pain" on the right end of the scale (10 cm). The patient will be asked to mark their current pain level on the line. They can also be asked to mark their maximum, minimum, and average pain. The examiner will score the VAS by measuring the distance in either centimeters (0 to 10) or millimeters (0 to 100) from the "no pain" anchor point.
Hand grip strength | up to five weeks
  Hand grip strength will be assessed by Hand grip dynamometer

CONTACTS AND LOCATIONS:
Overall Officials: Eman Em El halawany, Principal Investigator — Damanhour Teaching Hospital
Locations (1):
- Damanhour teaching hospital, Damanhūr, Egypt